CLINICAL TRIAL: NCT06797453
Title: Food Is Medicine Shared Medical Appointments for Weight Management: A Pilot Randomized Controlled Trial
Brief Title: Food is Medicine: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Ardmore Institute of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00117065
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Weight Loss
Keywords: Weight Management
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Completion of online Full Living Plate modules over eight weeks
  Interventions: Behavioral: Full Plate Living
- Intervention (Experimental): Attend shared medical visits over eight weeks and attend two cooking classes.
  Interventions: Behavioral: Shared Medical Visits

INTERVENTIONS:
Behavioral: Shared Medical Visits — Shared group medical visits over eight weeks and two cooking classes.
  Arms: Intervention
Behavioral: Full Plate Living — Online modules teaching how a high-fiber diet can lead to more energy, lower cholesterol, better blood sugar, and easier weight loss.
  Arms: Control

SUMMARY:
The goal of this study is to determine whether shared medical visits also called "group visits" would be beneficial for patients who are under weight management care.

As part of this study, participants will be asked to complete a survey to give the study team a better idea of their current health conditions and if this study will be good fit for them. Once the survey has been completed, participants will then be randomly assigned to one of two groups. Group one will include participation in shared medical visits over a period of eight weeks. In addition to the medical visits, this group will also include two cooking classes. Group two will be asked to complete online Full Living Plate modules. Participants will be asked to complete another survey at the end of the study.

DETAILED DESCRIPTION:
The purpose of this study is to have participants who are undergoing weight management attend new types of medical visits called "shared medical visits" and provide their feedback to the research staff. The shared medical visit or group visit is a new method of care delivery at Duke University Health System where patients with similar medical conditions have an appointment as a group with a provider. Patients can decide to share with the group or share privately with the provider team. Up to 50 people will take part in this study at Duke.

As part of this study, participants will be asked to complete a survey prior to starting the study to make sure that they are a good fit for the study.

Participants will be randomly assigned (like the flip of a coin) to one of two groups. Those placed in group one will have 4 group visit sessions that include 2 cooking demonstrations and those placed in group two will be asked to complete online Full Plate Living Modules. Both groups will receive the medically tailored groceries and can complete both the pre-survey and post-survey. Both groups will receive similar content, although only the individuals in the first option will have the opportunity to attend in-person group visit sessions. In-person sessions will be held at the Duke Integrative Medicine Center.

While on study, participants will receive medically tailored groceries delivered to their home every other week. Each delivery is about 70 servings of produce with possible additional grocery items.

If participants are unable to attend one of the group sessions while they are in the study, Telehealth group visits will be offered. However, this is not an alternative to an in-person class. This is being offered and approved by the study doctor on a case-by-case basis.

Participation in this study will last a total of eight weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients actively receiving care at the Duke Lifestyle and Weight Management Center (DLWMC)
2. Patients with obesity defined by BMI ≥30 kg/m2
3. Patients must live in Durham County
4. Patients age ≥18 years
5. Patients must be willing and able to consent to participating in 4 shared medical appointments with 10-13 other DLWMC patients over the course of 8 weeks
6. DLWMC provider must medically clear their participation in this program

Exclusion Criteria:

1. Patients with unstable medical or mental health condition, as deemed by their DLWMC medical provider (e.g., uncontrolled eating disorder, active severe major depression, gastrointestinal disease that would preclude consumption of a high fiber diet)
2. Patients who are pregnant or plan to become pregnant will be excluded, as change in weight will be a secondary outcome and patients may have specific dietary needs not covered by the content offered by this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Method (AIM) | 0 and 12 weeks
  "Acceptability" is defined as the perception among participants that a given treatment (food is medicine intervention with either group visits or online modules) is agreeable, palatable, or satisfactory. The AIM total score ranges from 1 to 20, where a higher score indicates greater acceptability.
Intervention Appropriateness Measure (IAM) | 0 and 12 weeks
  "Appropriateness" is defined as the perceived fit, relevance, or compatibility of the treatment (food is medicine intervention with either group visits or online modules) for the practice setting, provider, and participant; and/or perceived fit of the innovation to address obesity. The IAM total score ranges from 1 to 20, where a higher score indicates greater appropriateness.

SECONDARY OUTCOMES:
Fruit and Vegetable Consumption as measured by the 10-item Dietary Screener Questionnaire (DSQ) | 0 and 12 weeks
  The DSQ total score ranges from 0 to 100, where a higher score indicates greater fruit and vegetable consumption over the past month.
Number of participants with Nutrition Security | 0 and 12 weeks
  Nutrition security is defined as "consistent access, availability, and affordability of foods and beverages that promote well-being and prevent (and if needed, treat) disease."

CONTACTS AND LOCATIONS:
Overall Officials: Nia S Mitchell, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No